CLINICAL TRIAL: NCT03229954
Title: Intravenous Iron Isomaltoside 1000 (Monofer®) Compared With Oral Iron in the Treatment of Postgastrectomy Anemia: An Open-label Randomized Controlled Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2017-0149
Record Dates: First submitted 2017-07-23; First posted 2017-07-26 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Post Gastrectomy Anemia
MeSH Terms: interventions — iron isomaltoside 1000; Infusions, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IV iron (Monofer) group (Experimental): Iron isomaltoside(Monofer) will be injected intravenously and injection dose will be calculated using Ganzoni formula.
  Interventions: Drug: iron isomaltoside (Monofer) intravenous infusion
- Oral iron group (Active Comparator): Ferrous sulfate(Feroba-YOU) 160mg/day for 12 weeks will be taken per oral.
  Interventions: Drug: Ferrous sulfate(Feroba-YOU) per oral

INTERVENTIONS:
Drug: iron isomaltoside (Monofer) intravenous infusion — The investigational drug is a newest formulation of intravenous iron. The drug, iron isomaltoside (Monofer), will be infused one single high dose with infusion time more than 30 minutes (< 1,000 mg) or 60 minutes (≥ 1,000 mg). The dosage is determined using the Ganzoni formula and divided when the calculated dose exceeds 20 mg/kg.
  If the calculated dose exceeds 1,500 mg, the patient will be excluded from trial for patient safety.
  Arms: IV iron (Monofer) group
Drug: Ferrous sulfate(Feroba-YOU) per oral — 160 mg/day of ferrous sulfate (Feroba-YOU) will be taken per oral for 12 weeks.
  Arms: Oral iron group

SUMMARY:
Iron deficiency anemia is a common complication in patients who underwent gastrectomy and leads to a deterioration in patient's quality of life. Therefore iron supplementation is one of the important treatments in postgastrectomy patients.

Taking an oral iron is an option for iron supplementation, but the postgastrectomy patients has poor absorption of iron due to their anatomic change. Accordingly, intravenous iron supplementation has been emerged as another treatment option, but there are only a few studies to evaluate the efficacy of intravenous iron supplementation compared with oral iron in patients underwent gastrectomy.

Therefore, this study aims to evaluate the iron supplementation method as intravenous injection of iron isomaltoside compared with oral iron in the treatment of postgastrectomy anemia.

Gastric cancer patients who underwent curative gastrectomy more than 1 year ago and hemoglobin level lower than 11 g/dL will be included in this trial. After the registration, the patients will be randomly assigned to intravenous iron (n = 179) or oral iron groups (n = 179).

Calculated dose of iron isomaltoside using Ganzoni formula will be injected intravenously in intravenous iron group and 160 mg/day of ferrous sulfate for 12 weeks will be taken in oral iron group. Hemoglobin and iron profiles at baseline and weeks 2, 4, 8, and 12 and quality of life score at baseline and weeks 12 period will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥20 years of age
* Underwent gastrectomy for stage I or II of primary gastric adenocarcinoma
* Hb ≤11.0 g/dL at least one year after surgery
* Willingness to participate after signing informed consent

Exclusion Criteria:

* Calculated dosage using the Ganzoni formula >1,500 mg
* Any medical condition may have caused the patient to be unsuitable for the completion of the study or placed the patient at potential risk from being in the study
* Underwent chemotherapy or on chemotherapy
* Drug hypersensitivity to iron isomaltoside
* Active acute or chronic infections
* Known intolerance to oral iron treatment
* History of anemia due to extensive bleeding or causes other than iron deficiency
* Untreated vitamin B12 or folate deficiency
* Blood transfusion, Erythropoiesis stimulating agents(ESA), oral iron or intravenous iron treatment within 4 weeks prior to screening
* History of bone marrow suppression treatment, active Hepatitis B or C, HIV or hematologic disorder other than iron deficiency
* Iron overload, hematochromatosis or hemosiderosis
* Pregnancy or nursing
* Creatinine clearance rate using Cockcroft-Gault formula <30 mL/min
* Participation in any other clinical study within one month prior to screening

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Estimated)
Dates: Start 2017-08-28 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Hemoglobin at 2,4,8 and 12 weeks | at Baseline and weeks 2, 4, 8, and 12

SECONDARY OUTCOMES:
serum iron | at Baseline and weeks 2, 4, 8, and 12
serum ferritin | at Baseline and weeks 2, 4, 8, and 12
serum transferrin | at Baseline and weeks 2, 4, 8, and 12
transferrin saturation | at Baseline and weeks 2, 4, 8, and 12
QOL (quality of life) of the patients | at Baseline and weeks 2, 4, 8, and 12

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Yonsei University College of Medicine, Seoul, Korea, Seoul, South Korea